CLINICAL TRIAL: NCT06364085
Title: EPI-BOOST: Enhancing Epilepsy Management With Precision Deep Brain Stimulation
Brief Title: Enhancing Epilepsy Management With Precision Deep Brain Stimulation
Acronym: EPI-BOOST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Lutz Weise, Principal Investigator, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS2024
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Deep brain stimulation; DBS Programming
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participant Group (Experimental): Participants who meet eligibility criteria and provide informed consent.
  Interventions: Device: Neuromodulation programming

INTERVENTIONS:
Device: Neuromodulation programming — Participants will be brought in for their standard follow-up appointments at 4-weeks, 4-months, and 1-year post-surgery. In addition to the routine care, physiological data will be extracted from the implanted device and analyzed. The physiological data will be considered along with the standard epilepsy diary to assess epileptic burden and inform device programming.
  Quality of life will be measured with a series of standard questionnaires pre-surgery and at the 1-year follow-up.

SUMMARY:
The goal of this study is to evaluate the effectiveness of objective neural response feedback on deep brain stimulation (DBS) programming for drug-resistant epilepsy in a prospective observational cohort study.

DETAILED DESCRIPTION:
Aim 1: To objectively monitor epilepsy burden with the provided sensing capabilities of the DBS leads by quantifying the association between neuronal activity and seizure frequency

Aim 2: To use the neuronal activity to inform programming of DBS for patients with epilepsy, and assess the impact on patient and caregiver quality of life and hospital costs.

Epilepsy is a neurological disorder characterized by recurrent, unprovoked seizures that affects millions of individuals worldwide and poses a significant burden on their quality of life. Despite considerable advancements in treatment strategies, approximately one-third of patients are considered to have drug-resistant epilepsy. Patients with drug-resistant epilepsy frequently visit the emergency room, are hospitalized regularly, and have many seizure-related injuries. Deep brain stimulation (DBS) offers a unique treatment option by delivering precise electrical pulses with surgically implanted electrodes to the specific brain regions responsible for seizures, disrupting the seizure pathways. Long-term favorable findings showing significant seizure reduction at five-year post-implantation for patients who otherwise have no treatment options have convinced many centers to incorporate DBS into their healthcare practise.

For assessing the treatment response in epilepsy, healthcare providers are dependent on patient-reported seizure diaries. Recent research in DBS has focused on the biological implications of neuronal recordings through the implanted electrodes. These signals offer objective insight into brain activity, specifically epileptic burden, and offers potentially predictive capabilities. Current research focuses on whether the sensing capabilities of DBS can provide reliable seizure burden detection, and whether this can be achieved with less demand on the patient.

In this prospective observational cohort study, the researchers aim to improve the impact of DBS treatment on the seizure burden and quality of life of patients diagnosed with drug-resistant epilepsy in Atlantic Canada. This will be done by investigating the neural activity underlying epileptic events as a representation of epileptic burden, affording the opportunity to tailor DBS interventions with more precision and efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualifying for deep brain stimulation on the basis of drug-resistant epilepsy
* Informed consent

Exclusion Criteria:

* Lack of consent
* Electrical or other devices that preclude the performance of an MRI for pre-operative imaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Seizure reduction | Change from baseline versus Month 12
  The number of seizures experienced by patients will be assessed by the number of seizures recorded by patients and their caregivers in seizure diaries and described as absolute seizure reduction.

SECONDARY OUTCOMES:
Change in disease score on Patient Weighted Quality Of Life In Epilepsy | Twelve months
  Assessment of therapeutic effects using Patient Weighted Quality Of Life In Epilepsy, a 10-question survey completed by patients to assess quality of life, where a higher score is associated with a more positive quality of life.
Change in depression score on Neurological Disorders Depression Inventory in Epilepsy | Twelve months
  Assessment of therapeutic effects using Neurological Disorders Depression Inventory in Epilepsy, a 6-question survey to assess depression. A higher score is associated with more severe depression.
Change in anxiety score on Anxiety General Anxiety Disorder-7 | Twelve months
  Assessment of therapeutic effects using Anxiety General Anxiety Disorder-7, a 7-question survey to assess anxiety. A higher score is associated with more severe anxiety, and a lower score is associated with minimal anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Weise, MD, PhD, Principal Investigator — Dalhousie University
Locations (1):
- Queen Elizabeth Health Science Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No